CLINICAL TRIAL: NCT04910048
Title: Impact of a Preoperative Patient Optimization Program on Preoperative Health, Eligibility, and Clinical & Patient-Reported Outcomes in Total Joint Arthroplasty
Brief Title: Impact of a POPOP on Preoperative Health, Eligibility, and Clinical & Patient-Reported Outcomes in TJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262790
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Avascular Necrosis; Rheumatoid Arthritis
Keywords: Total joint arthroplasty; Hip arthroplasty; Knee arthroplasty; Surgical ineligibility; Obesity; Patient Reported Outcome Measures; TJA; THA; TKA; PROMs; BMI; HbA1c
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteonecrosis; Arthritis, Rheumatoid; Obesity | interventions — POPOP; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two group randomized control trial comparing the intervention (POPOP) and standard of care (SOC).
Masking Description: Due to the nature of the interventions, masking or blinded participation is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): The first arm consists of UAMS standard of care (SOC), including providing a brochure with information (contact information, brief educational information) for the patient to consult with a nutritionist to help with self-directed weight loss.
  Interventions: Other: SOC (standard of care)
- Intervention (POPOP) (Experimental): The second arm is a specified 2-month POPOP focused on weight loss administered by the external partner, 20Lighter. The program includes customized meal plans; vitamin, mineral and nutritional supplementation; and daily engagement via a smartphone app with a 20Lighter health care provider. Video conferencing appointments will occur approximately every 3 weeks. The program does not require any exercise or physical engagement but does necessitate that patients have a smartphone or tablet with Bluetooth capability, cell signal or WIFI connection. During the first 40 days the customized meal plans are adhered to, then from days 41-60 patients will transition back to a normal dietary lifestyle via a customized plan based on considerations including, food preferences, physical engagement and height. Patients who achieve a BMI below 40.0 before the end of the 60 day program may be seen sooner than 90d for follow-up appointment in the UAMS clinic.
  Interventions: Other: POPOP (preoperative patient optimization program)

INTERVENTIONS:
Other: POPOP (preoperative patient optimization program) — A 2 month structured program focused on reduction of BMI, body weight, visceral fat, body fat and improvement of lean body mass and intracellular fluid.
  Other Names: 20Lighter
  Arms: Intervention (POPOP)
Other: SOC (standard of care) — Referral to a dietician for two months of self-directed weight loss
  Arms: Standard of Care

SUMMARY:
In this pilot study, we will test the hypothesis that a POPOP for currently ineligible UAMS orthopedic surgery patients wanting hip or knee replacement improves markers of preoperative health, ability to reach a BMI threshold <40 kg/m2 required for surgical eligibility, and postoperative outcomes versus SOC.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be screened to determine eligibility for study entry. Patients who meet eligibility criteria will be randomized into one of two groups: Standard of Care or the POPOP (20Lighter).

ELIGIBILITY:
Inclusion Criteria:

* End-stage knee or hip osteoarthritis, avascular necrosis, or rheumatoid arthritis with recommended primary, unilateral total joint arthroplasty by orthopaedic surgeons at the University of Arkansas for Medical Sciences (Jeffrey Stambough, Dr. C. Lowry Barnes, Dr. Simon Mears, and Dr. Benjamin Stronach)
* BMI between 41.00-48.00 kg/m2 at time of enrollment
* Over the age of 18 years
* Would consider undergoing a total joint arthroplasty if eligible
* Owns a smartphone or tablet with Bluetooth capability, cell signal or WIFI connection
* Willing to comply with the requirements of the study and provide informed consent prior to enrollment.

Exclusion Criteria:

* Patients with a BMI less than 41.00 or greater than 48.00
* Pregnancy
* Breastfeeding
* History of a major organ transplant or other health issue requiring immunosuppressant drugs
* Strict vegetarian diet
* Diagnosis of and/or are taking medication for psychiatric conditions including schizophrenia, bipolar disorder or manic depression
* Patients scheduled for, or those who have previously undergone, bariatric surgery
* Patients unable to understand and speak English
* Patients requiring a revision or bilateral TJA
* Patients unwilling or unable to use a bluetooth-enabled smartphone with cell service or home internet access
* Incarceration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Change of pre-operative BMI | Approximately 70-110 days from study enrollment
  Assessment of mean change in BMI (Body Mass Index, kg/m2) between the date of enrollment to follow-up visit to occur between days 70-110

SECONDARY OUTCOMES:
Pre-operative health & nutritional status as assessed by change of red blood cell count | Approximately 70-110 days from study enrollment
  Change of values in red blood cells as assessed by (Complete Blood Count) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of white blood cell count | Approximately 70-110 days from study enrollment
  Change of values in white blood cells as assessed by CBC (Complete Blood Count) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of platelet count | Approximately 70-110 days from study enrollment
  Change of values in platelets as assessed by CBC (Complete Blood Count) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of albumin | Approximately 70-110 days from study enrollment
  Change of values in Albumin as assessed by CMP (Comprehensive Metabolic Panel) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of ALT (alanine aminotransferase) | Approximately 70-110 days from study enrollment
  Change of values in ALT (alanine aminotransferase) as assessed by CMP (Comprehensive Metabolic Panel) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of AST (aspartate aminotransferase) | Approximately 70-110 days from study enrollment
  Change of values in AST (aspartate aminotransferase) as assessed by CMP (Comprehensive Metabolic Panel) between the date of enrollment to follow-up visit to occur between days 70-110
Pre-operative health & nutritional status as assessed by change of BUN (blood urea nitrogen) | Approximately 70-110 days from study enrollment
  Change of values in BUN (blood urea nitrogen) as assessed by CMP (Comprehensive Metabolic Panel) between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative health & nutritional status as assessed by Creatinine | Approximately 70-110 days from study enrollment
  Change of values in Creatinine as assessed by CMP (Comprehensive Metabolic Panel) between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative type 2 diabetes as assessed by HbA1c (Hemaglobin A1c) laboratory test values | Approximately 70-110 days from study enrollment
  Assessment of change in HbA1c (Hemaglobin A1c) between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative inflammation as assessed by CRP (C-Reactive Protein) laboratory test values | Approximately 70-110 days from study enrollment
  Assessment of change in CRP (C-Reactive Protein) between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative PROMs (Knee Replacement) | Approximately 70-110 days from study enrollment
  Assessment of change in the patient reported outcomes survey KOOS Jr, knee replacement patients between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative PROMs (Hip Replacement) | Approximately 70-110 days from study enrollment
  Assessment of change in the patient reported outcomes survey HOOS Jr, hip replacement patients between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative PROMIS Pain Interference | Approximately 70-110 days from study enrollment
  Assessment of change in PROMIS Pain Interference patient reported outcome instrument between the date of enrollment to follow-up visit to occur between days 70-110
Change of pre-operative PROMIS Physical Function | Approximately 70-110 days from study enrollment
  Assessment of change in PROMIS Physical Function patient reported outcome instrument between the date of enrollment to follow-up visit to occur between days 70-110

OTHER OUTCOMES:
Percentage of patients converting from ineligible to eligible status | Approximately 70-110 days from study enrollment
  Assessment of the percentage of patients achieving a BMI of 40.0 kg/m2 or less in each treatment group
Percentage of patients who proceed to TJA | Approximately 110-120 days from study enrollment
  Assessment of the percentage of patients that undergo TJA in each treatment group
Change of PROMs in the 6-weeks after knee replacement | Approximately 180 days from study enrollment (or 6 weeks after TJA)
  Assessment of change in the patient reported outcomes survey KOOS Jr, for patients undergoing knee replacement
Change of PROMs in the 6-weeks after hip replacement | Approximately 180 days from study enrollment (or 6 weeks after TJA)
  Assessment of change in the patient reported outcomes survey HOOS Jr, for patients undergoing hip replacement
Change of PROMIS Pain Interference in the 6-weeks after joint replacement | Approximately 180 days from study enrollment (or 6 weeks after TJA)
  Assessment of change in PROMIS Pain Interference patient reported outcome instrument
Change of PROMIS Physical Function in the 6-weeks after joint replacement | Approximately 180 days from study enrollment (or 6 weeks after TJA)
  Assessment of change in PROMIS Physical Function patient reported outcome instrument
All-cause complication rate at 30-days post TJA | Approximately 160 days from study enrollment (or 30 days after TJA)
  Rate of surgical complications requiring hospital readmission, ER or acute care visit in 30 days after TJA
All-cause complication rate at 60-days post TJA | Approximately 190 days from study enrollment (or 60 days after TJA)
  Rate of surgical complications requiring hospital readmission, ER or acute care visit in 60 days after TJA
All-cause complication rate at 90-days post TJA | Approximately 220 days from study enrollment (or 90 days after TJA)
  Rate of surgical complications requiring hospital readmission, ER or acute care visit in 90 days after TJA

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Stambough, MD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS Orthopaedic Clinic - Shackleford, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Statistics based on aggregated de-identified data will be assessed, and disseminated at industry conferences and peer-reviewed publication.

REFERENCES:
- [Background] Bolognesi MP, Marchant MH Jr, Viens NA, Cook C, Pietrobon R, Vail TP. The impact of diabetes on perioperative patient outcomes after total hip and total knee arthroplasty in the United States. J Arthroplasty. 2008 Sep;23(6 Suppl 1):92-8. doi: 10.1016/j.arth.2008.05.012. PMID 18722309
- [Background] Boyce L, Prasad A, Barrett M, Dawson-Bowling S, Millington S, Hanna SA, Achan P. The outcomes of total knee arthroplasty in morbidly obese patients: a systematic review of the literature. Arch Orthop Trauma Surg. 2019 Apr;139(4):553-560. doi: 10.1007/s00402-019-03127-5. Epub 2019 Feb 16. PMID 30778723
- [Background] Gerlach E, Selley R, Johnson D, Nicolay R, Versteeg G, Plantz M, Tjong V, Terry M. Patient-Reported Outcomes Measurement Information System Validation in Hip Arthroscopy: A Shift Towards Reducing Survey Burden. Cureus. 2021 Feb 10;13(2):e13265. doi: 10.7759/cureus.13265. PMID 33728201
- [Background] Goodman SM, Mehta BY, Mandl LA, Szymonifka JD, Finik J, Figgie MP, Navarro-Millan IY, Bostrom MP, Parks ML, Padgett DE, McLawhorn AS, Antao VC, Yates AJ, Springer BD, Lyman SL, Singh JA. Validation of the Hip Disability and Osteoarthritis Outcome Score and Knee Injury and Osteoarthritis Outcome Score Pain and Function Subscales for Use in Total Hip Replacement and Total Knee Replacement Clinical Trials. J Arthroplasty. 2020 May;35(5):1200-1207.e4. doi: 10.1016/j.arth.2019.12.038. Epub 2019 Dec 27. PMID 31952945
- [Background] Harold RE, Butler BA, Delagrammaticas D, Sullivan R, Stover M, Manning DW. Patient-Reported Outcomes Measurement Information System Correlates With Modified Harris Hip Score in Total Hip Arthroplasty. Orthopedics. 2021 Jan 1;44(1):e19-e25. doi: 10.3928/01477447-20201202-02. Epub 2020 Dec 7. PMID 33284982
- [Background] Horn ME, Reinke EK, Couce LJ, Reeve BB, Ledbetter L, George SZ. Reporting and utilization of Patient-Reported Outcomes Measurement Information System(R) (PROMIS(R)) measures in orthopedic research and practice: a systematic review. J Orthop Surg Res. 2020 Nov 23;15(1):553. doi: 10.1186/s13018-020-02068-9. PMID 33228699
- [Background] Keeney BJ, Austin DC, Jevsevar DS. Preoperative Weight Loss for Morbidly Obese Patients Undergoing Total Knee Arthroplasty: Determining the Necessary Amount. J Bone Joint Surg Am. 2019 Aug 21;101(16):1440-1450. doi: 10.2106/JBJS.18.01136. PMID 31436651
- [Background] Lingamfelter M, Orozco FR, Beck CN, Harrer MF, Post ZD, Ong AC, Ponzio DY. Nutritional Counseling Program for Morbidly Obese Patients Enables Weight Optimization for Safe Total Joint Arthroplasty. Orthopedics. 2020 Jul 1;43(4):e316-e322. doi: 10.3928/01477447-20200521-08. Epub 2020 Jun 5. PMID 32501522
- [Background] Shaka H, Ojemolon PE. Impact of Obesity on Outcomes of Patients With Hip Osteoarthritis Who Underwent Hip Arthroplasty. Cureus. 2020 Oct 10;12(10):e10876. doi: 10.7759/cureus.10876. PMID 33178529
- [Background] Shapiro JA, Narayanan AS, Taylor PR, Olcott CW, Del Gaizo DJ. Fate of the Morbidly Obese Patient Who Is Denied Total Joint Arthroplasty. J Arthroplasty. 2020 Jun;35(6S):S124-S128. doi: 10.1016/j.arth.2020.01.071. Epub 2020 Feb 4. PMID 32088050